CLINICAL TRIAL: NCT06065813
Title: The Efficacy and Safety of Neoadjuvant Triprizumab and Radiotherapy in Operable Patients With Stage IIB-IIIA Non-small Cell Lung Cancer
Brief Title: Neoadjuvant Triprizumab and Radiotherapy in Operable Patients With Stage IIA-IIIA Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Principal Investigator, Buhai Wang, Director, Northern Jiangsu People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LC-001
Record Dates: First submitted 2023-09-06; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Non-small Cell Lung Cancer; Neoadjuvant Therapy; Radiotherapy; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab (Experimental)
  Interventions: Drug: Toripalimab; Radiation: Conventional segmental radiotherapy; Other: opreation

INTERVENTIONS:
Drug: Toripalimab — 200 mg Toripalimab intravenously every 3 weeks 3 doses of Toripalimab before operation 14 doses of Toripalimab 30 days after operation
  Other Names: JS001
Radiation: Conventional segmental radiotherapy — the does of radiation will be 40-45Gy. The day of the first dose of Toripalimab and the first day of radiation must be the same day.
Other: opreation — The operable patients will accept radical operated in 28-42 days after the third dose of Toripalimab

SUMMARY:
Neoadjuvant Triprizumab and Radiotherapy in Operable Patients With Stage IIA-IIIA Non-small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients must volunteer participating in clinical trial; patients fully understand and sign the Informed Consent Form (ICF)
* 18 ~ 70 years old, gender not limited
* Histologically confirmed resectable stage IIA-IIIA NSCLC without prior treatment
* Patients must have at least one "target" lesion" to be used to assess response on this protocol as defined by RECIST 1.1
* Agree to provide PD-L1 immune tissue sections and corresponding pathology reports for biomarker evaluation (Tumor tissue samples must be fresh or archived samples obtained within 3 months before enrollment
* Have a performance status of 0 or 1 on the ECOG Performance Scale
* Good organ function: ANC ≥ 1500/μL; PLT ≥ 100000/μL; HB ≥ 10.0g/dL; CR ≤ 1.5 × ULN or CrCl ≥ 60 mL/min (Use Cock-Gault formula); TB ≤ 1.5 × ULN (For patients with total bilirubin levels > 1.5 × ULN, direct bilirubin is within normal limits); AST and ALT ≤ 2.5 × ULN; TSH is within normal limits. Note: If TSH is not within the normal range at baseline, if T3 and free T4 are within the normal range, then the patient can still meet the inclusion criteria. IN、RPT、APTT≤1.5×ULN
* Patients must volunteer and be able to follow research plan visits, treatment plans, laboratory tests, and other research procedures
* According to the surgeon's assessment, the total lung function can withstand the proposed lung resection
* Within 3 days before medication，the serum of fertile woman must be tested by hcg，and the result is negative. Fertile women can use high effective method for contraception in the duration of clinical trail and 180 days after last Administration

Exclusion Criteria:

* Locally advanced unresectable or metastatic disease
* Non-small small lung cancer (NSCLC) involving the upper sulcus，large cell neuroendocrine cancer (LCNEC), sarcomatoid tumor
* Patients with known EGFR mutations or ALK translocations, non-squamous carcinoma patients need to know the status of EGFR and ALK mutations
* Early NSCLC with prior systemic anticancer therapy, including experimental drug therapy
* Have a history of (non-infectious) pneumonia / interstitial lung disease requiring steroid therapy, or currently have pneumonia / interstitial lung disease requiring steroid therapy
* Known history of active tuberculosis
* Known to have active infection requiring systemic treatment
* known or suspected autoimmune diseases or immunodeficiency, except: patients with a history of hypothyroidism who do not require hormone therapy or are receiving physiological dose hormone replacement therapy; patients with stable type 1 diabetes whose blood glucose is controlled
* Active hepatitis B or C
* Has a known history of Human Immunodeficiency Virus (HIV) .
* Received live vaccine treatment within 30 days before drug administration; but inactivated viral vaccine for seasonal influenza is allowed
* Peripheral neuropathy ≥ grade 2
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Overly sensitive reaction to other monoclonal antibodies
* Have a history of severe allergies to pemetrexed, paclitaxel or docetaxel, cisplatin, carboplatin or their preventive medicine
* Known to have serious or uncontrolled underlying disease
* According to the investigator's judgment, the patient has a history or current evidence of any disease, treatment or laboratory abnormality that may confuse the test results, interfere with the participant's participation in the full trial, or not in the best interest of the participant to participate in the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response rates | 42months
  Major pathological response rates assessed by independent center pathology
Event-free survival | 42months
  The time from the beginning of enrollment to the occurrence of any events, including death, disease progression, change of chemotherapy regimen, change of chemotherapy, addition of other treatments, the occurrence of fatal or intolerant side effects and other events

SECONDARY OUTCOMES:
Overall survival | 42 months
  Kaplan-Meier median estimates and curves will be used to describe OS survival functions
Pathologic complete response (pCR) rates | 42months
  Pathologic complete response (pCR) rate is defined as the number of randomized participants with absence of residual tumor in lung and lymph nodes as evaluated by blinded independent pathological review.
Disease-free survival | 42 months
  Some time until the tumor recurs or die for various reasons
Number of Participants Experiencing Adverse Events (AEs) and serious adverse events (SAEs) | 42 months
  Adverse events are defined as any adverse medical events that occur in the participants taking the drugs and do not necessarily have a causal relationship with the treatment. AEs/SAEs were evaluated using NCI-CTCAE v5.0

OTHER OUTCOMES:
Biomarkers | 42 months
  PD-L1 expression of tissue specimens、TMB、WES and changes of ctDNA in peripheral blood

CONTACTS AND LOCATIONS:
Locations (1):
- People's hospital of northern jiangsu, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No